CLINICAL TRIAL: NCT00540072
Title: Study of Cidecin™ (Daptomycin) to Rocephin® (Ceftriaxone) in the Treatment of Moderate to Severe Community-Acquired Acute Bacterial Pneumonia Due to S. Pneumoniae
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DAP-CAP-00-08
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Pneumonia, Bacterial
Keywords: Moderate to Severe Community-Acquired Acute Bacterial Pneumonia Due to S. Pneumoniae
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — Daptomycin

INTERVENTIONS:
Drug: daptomycin

SUMMARY:
A COMPARASON OF CIDECIN™ (DAPTOMYCIN) TO ROCEPHIN® (CEFTRIAXONE) IN THE TREATMENT OF MODERATE TO SEVERE COMMUNITY-ACQUIRED ACUTE BACTERIAL PNEUMONIA DUE TO S. PNEUMONIAE

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent.
2. Adults, 18 years of age or older of either gender and of any race weighing up to 150 kg. Female patients of childbearing potential MUST be nonpregnant (confirmed by negative serum pregnancy test), nonlactating, and must be willing to practice reliable birth control measures during and for at least 30 days after treatment with study drug(s).
3. Have a new pulmonary infiltrate on chest radiograph.
4. Exhibit at least two of the following clinical symptoms of pneumonia on history or physical:

   * Cough
   * Production of purulent sputum or change in character of sputum
   * Auscultatory findings on pulmonary examination of rales and/or evidence of pulmonary consolidation (dullness to percussion, bronchial breath sounds, or egophony)
   * Dyspnea or tachypnea
   * Documented fever, defined as body temperature >38.0 ºC (100.4 ºF) taken orally; >38.5 ºC (101.2 ºF) tympanically; or >39.0 ºC (102.2 ºF) rectally or hypothermia, defined as core body temperature of <35.0 ºC (95.0 ºF)
   * An elevated total peripheral white blood cell count (WBC >10,000/mm3); or >15% immature neutrophils (bands), regardless of total peripheral white count; or leukopenia with total WBC <4500/mm3.
   * Hypoxemia with a PO2 < 60 mmHg (on room air) or O2 saturation <90% on room air
5. Pneumonia which requires hospitalization and intravenous therapy for at least 5 days.
6. Willingness to participate in this study and to complete all follow-up assessments.

Exclusion Criteria:

1. Patients with Grade V pneumonia (based on Fine Score; Attachment 8).
2. Patients in respiratory failure or incipient respiratory failure if the patient is not a candidate for mechanical ventilation (for any reason).
3. Any of the following pulmonary conditions that may preclude interpretation of study results:

   * Cystic fibrosis
   * Primary lung cancer or another malignancy metastatic to the lungs
   * Known bronchial obstruction or a history of post-obstructive pneumonia
   * Known or suspected active tuberculosis.
4. Severe shock (systolic blood pressure <90 mm Hg for >30 minutes not corrected by fluid bolus).
5. Clinical evidence of bacterial meningitis (based on lumbar puncture results).
6. Severe renal impairment (calculated creatinine clearance <30 mL/min).
7. Moribund clinical condition: high likelihood of death during the first 48 hours.
8. If HIV positive, known CD4 counts <200/mm3 or evidence of Pneumocystis carinii pneumonia.
9. Inability to tolerate ceftriaxone or history of allergy to beta-lactam antibiotics (history of rash alone will not exclude a patient).
10. Any individual previously treated with a potentially effective anti-infective agent for > 24 hours (or one dosing day) within 72 hours of enrollment, or prior treatment with any investigational drug (including experimental biologic agents) in previous 30 days or prior therapy with daptomycin.
11. Patients who must continue HMG-CoA reductase inhibitor therapy (e.g., simvastatin, lovastatin, etc.) during the study treatment period.
12. Anticipation that a second non-protocol systemic antibiotic will be required.
13. Induction chemotherapy within 2 weeks prior to enrollment (or exogenous therapies which are anticipated to result in PMN counts of <200 mm3 during Treatment Phase), or patients with severe neutropenia (<200 PMN cells/mm3).
14. Patients considered unreliable to return for visits or to comply with study procedures.
15. Progressive neoplastic disease (Note: patients with malignancies in remission are eligible).
16. Women who are pregnant or nursing/lactating.
17. Patients presenting with nosocomial pneumonia (i.e., <14 days after discharge from a skilled nursing facility or hospital with an initial hospitalization of >=3 days duration).
18. Clinical suspicion of Legionella pneumonia.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2001-07-30 (Actual); Primary Completion 2002-02-27 (Actual); Study Completion 2002-02-27 (Actual)

REFERENCES:
- [Result] Pertel PE, Bernardo P, Fogarty C, Matthews P, Northland R, Benvenuto M, Thorne GM, Luperchio SA, Arbeit RD, Alder J. Effects of prior effective therapy on the efficacy of daptomycin and ceftriaxone for the treatment of community-acquired pneumonia. Clin Infect Dis. 2008 Apr 15;46(8):1142-51. doi: 10.1086/533441. PMID 18444848